CLINICAL TRIAL: NCT06442293
Title: An Evaluation of the Safety and Tolerability of 2 Dietary Supplement Beverages Designed to Maintain Normal Blood Pressure in Normal, Healthy Individuals.
Brief Title: Safety and Tolerability of 2 Dietary Supplement Beverages Designed to Maintain Healthy Blood Pressure.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202401CT
Record Dates: First submitted 2024-04-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Safety Issues; Tolerance

STUDY DESIGN:
Intervention Model Description: single blind, placebo controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): a placebo (microcrystalline cellulose) identical in size, shape and color to the treatment
  Interventions: Dietary Supplement: Placebo
- Circulatory Beverage - low dose (Experimental): A beverage containing natural ingredients at a low dose
  Interventions: Dietary Supplement: Treatment 1
- Circulatory Beverage - medium dose (Experimental): A beverage containing natural ingredients at a medium dose
  Interventions: Dietary Supplement: Treatment 1
- Circulatory Beverage - high dose (Experimental): A beverage containing natural ingredients at a high dose
  Interventions: Dietary Supplement: Treatment 1
- TCM Beverage - low dose (Experimental): A traditional Chinese medicine-based beverage containing natural ingredients at a low dose
  Interventions: Dietary Supplement: Treatment 2
- TCM Beverage - high dose (Experimental): A traditional Chinese medicine-based beverage containing natural ingredients at a high dose
  Interventions: Dietary Supplement: Treatment 2

INTERVENTIONS:
Dietary Supplement: Treatment 1 — A dietary supplement containing beet root extract, arginine and citrulline
  Arms: Circulatory Beverage - high dose; Circulatory Beverage - low dose; Circulatory Beverage - medium dose
Dietary Supplement: Treatment 2 — A traditional Chinese medicine (TCM)-based dietary supplement containing chrysanthemum extract and eucommia bark extract
  Arms: TCM Beverage - high dose; TCM Beverage - low dose
Dietary Supplement: Placebo — a placebo supplement that is similar in appearance to treatment 1
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and tolerability of two distinct dietary supplement beverage formulations designed to maintain normal blood pressure. In this study, safety and tolerability will be assessed among otherwise healthy, normotensive individuals.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety of 2 dietary supplement beverage formulations in healthy, normotensive individuals. The study period will be 29 days in length, during which we will monitor and catalogue the blood pressure (BP), heart rate (HR), comprehensive metabolic panel (CMP), complete blood count (CBC), as well as self-reported side effects of all subjects on a daily basis. Note that each beverage will be evaluated at multiple doses: Beverage 1 will be monitored at a low, medium and high dose, where the medium and high dose is quantitatively twice (2X) and thrice (3X) the low dose (1X), respectively. Similarly, we will evaluate Beverage 2 at a low dose and high dose where the high dose is quantitatively twice (2X) of the low dose (1X). A placebo treatment will also be incorporated into this study as well. As such, there will be 6 groups in this study. Three subjects will be assigned to each treatment group for a total of 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

* You are male or female between the ages of 18 and 50 (inclusive)
* You are in generally good health and taking no medications known to treat or affect blood pressure (e.g., angiotensin converting enzyme (ACE) inhibitors, calcium channel blockers, diuretics)
* You have a Body Mass Index of 18.5 to 30.0
* You have a resting blood pressure of systolic blood pressure (SBP) of 90 - 120 mm Hg and a diastolic blood pressure (DBP) 60 - 80 mm Hg
* You are comfortable reading and speaking in English
* You are fully able and willing to comply with the requirements of the study
* You are fully able and willing to keep scheduled appointments
* You have no known food allergies or intolerances
* Female individuals will be asked to complete a pregnancy screening test.

Exclusion Criteria:

* You are pregnant, attempting to become pregnant, or are currently lactating
* You currently use prescription or over-the-counter medications that may interfere with absorption of the test supplement or confound results (e.g., thiazide and loop diuretics for hypertension, corticosteroids)
* You have clinically important gastrointestinal, renal, hepatic, cardiac, pulmonary, pancreatic, neurologic or biliary disorders or conditions. Individuals with type 1 or type 2 diabetes will be excluded from the study
* You have illnesses or other medical conditions that will prevent or interfere with giving an informed consent, or with participation in the study.
* You have scheduling difficulties or lack of transportation that will prevent or interfere with their ability to attend all the necessary study visits.
* You have participated as a subject in any other clinical study within 30 days of the screening visit.
* You have a history of alcohol abuse or other substance abuse within the previous 2 years.
* You are currently using tobacco products including chewing tobacco and cigarettes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Aggregate Adverse Symptom Score | 4 weeks
  An assessment of adverse symptoms categorized as either respiratory, cardiovascular, neurological or gastrointestinal. If symptoms present, they are rated on a scale from 1 to 10, with indicating very mild symptoms and 10 indicating very severe symptoms.

SECONDARY OUTCOMES:
Blood pressure assessment | 4 weeks
  An assessment of subjects' blood pressure throughout the 4-week study period.
Heart rate monitoring | 4 weeks
  An assessment of subjects' heart rate throughout the 4-week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levy, PhD, Principal Investigator — USANA Health Sciences
Locations (1):
- USANA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No